CLINICAL TRIAL: NCT05862415
Title: Impact of Two Types of Concurrent Training for Optimal Physiological and Physical Benefits in Middle-Aged Adults: a Randomized Controlled Trial
Brief Title: Concurrent Training for Optimal Physiological and Physical Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monira Aldhahi (Other)
Responsible Party: Sponsor-Investigator, Monira Aldhahi, Assistant professor, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 198511
Record Dates: First submitted 2023-04-25; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Healthy; Physical Inactivity
Keywords: Anaerobic work; Endurance; Aerobic training; Concurrent Training
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strength+aerobic group (SAG) (Active Comparator): All training sessions began with a 5- to 7-minute warm- up (consisting low-intensity walking and running, and dynamic mobility exercises) and active recovery of 4- to 5-minute (based on stretching and relaxation exercises). Sessions lasted approximately 50 minutes (warm-up and cold down included), with an overall weekly volume of 105-120 minutes.
  The circular training method was used in the resistance training phase. During the aerobic training phase, a series of movements from moderate intensity to vigorous intensity was performed.
  The RT lasted approximately 20-25 min per session and included two sets of 8-20 repetitions, with a rest interval of 1-2 min. The resistance training program was performed using the circuit training method in which two or three sets were performed. The RT exercises included: squat, barbell bent-over row, overhead press, plank, lateral pull down, triceps push down, barbell curl, leg extension, leg curl, lunge, barbell bench press, crunches etc.
  Interventions: Other: therapeutic Exercise
- aerobic+strength group (ASG) (Experimental): Similar to the active comparator group, but the order of the training reverse.
  Interventions: Other: therapeutic Exercise

INTERVENTIONS:
Other: therapeutic Exercise — The circular training method was used in the resistance training phase. During the aerobic training phase, a series of movements from moderate intensity to vigorous intensity was performed. The step loading periodization principle was taken into account in both resistance training and aerobic exercises.
  The RT lasted approximately 20-25 min per session and included two sets of 8-20 repetitions, with a rest interval of 1-2 min. The RT exercises included: squat, barbell bent-over row, overhead press, plank, lateral pull down, triceps push down, barbell curl, leg extension, leg curl, lunge, barbell bench press, crunches etc.
  For the aerobic training: Intensity was established between 50-65% and 80-85% of HRmax for both groups (SAG and ASG). Aerobic training includes walking and running periods and was carried out on a 400 m outdoor track. In periodization, especially 1st-4th.

SUMMARY:
It is widely accepted that aerobic exercise and strengthen training are the core components of most workout programs. However, there is no clear consensus on whether the order in which the exercises are performed impacts their effectiveness. Therefore, the overarching aim of the study is to understand the optimal order of two types of concurrent training program for 13 weeks by comparing the effectiveness of the training on body composition, predicated maximal oxygen uptake (MaxVO2), dynamic respiratory parameters, and muscle strength in healthy middle-aged people. Methods:Thirty-three moderately-active middle-aged and healthy participants were randomly assigned to the strength+aerobic group (SAG, n = 16) and aerobic+strength group (ASG, n = 17). Body composition, aerobic endurance, respiratory parameters and upper and lower strength were assessed before (pre-test) and after (post-test) a 13-week intervention. The chi-square test and the independent t-test will be used to compare sociodemographic variables between the groups. A 2 x 2 analysis of variance (ANOVA) with repeated measures (group x measurement) will be conducted.

This study will enhance our understanding of the concurrent training effect on muscle composition and strength. These training programs allow for reducing the duration of the training, which can be an important factor in making adults more willing to participate in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* middle-aged adults ( over the age of 40)
* No history of cardiovascular or neuromuscular disorders
* not having orthopedic disorder or neurologic disorders.

Exclusion Criteria:

* adults using artificial prosthesis
* participation in any structured training program
* any disease that precludes exercise or necessitates special care (for example, coronary artery disease, thrombosis, moderate or severe bone disease, and lung or renal disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Body fat % | 10 min
  To measure the BF%, a bioelectrical impedance analysis was used. The participants will be instructed to stand barefoot on the bioelectrical impedance analysis devices (seca mBCA 515, Hamburg, Germany).The device measures the body composition and includes a platform with handrails and electrodes that measure the impedance passed through the pairs of hands and feet while standing. Impedance was measured over 75 s with a current of 100 μA at a frequency range between 1 kHz and 1000 kHz and a capacity of 360 kg. Waist circumference measurement at the umbilicus and level physical activity level were inputted to indirectly estimate the body composition.
Predicated maximal oxygen uptake (MaxVO2) | 1 day
  1-mile walk-run performance test was used. The aim of this test is to cover a distance of one mile in the shortest possible time. Participants can alternate between walking and running as desired; however, they should be encouraged to cover the distance as quickly as feasible. The time elapsed to cover a mile distance, measured in minutes and seconds. During the testing and recovery the heart rate of the participants was monitored with a heart rate sensor (Polar Verity Sense; Kempele, Finland). Polar Verity Sense can be connected to a sports watch or app via Bluetooth®, ANT+, and internal memory to instantly track your training or view the data after training. As a result, the participant's time for completing the 1-mile test was tracked using a smart phone GPS system. The validity of the device has previously been reported previously[27]. The participants' MaxVO2 values were calculated using the formulas below.
Forced Vital Capacity (FVC) | 1 day
  a spirometer device (Minispir®, PC-based Spirometer with Oximetry option, Italy) will be used to measure the Forced Vital Capacity (FVC), Forced Expiratory Volume in One Second (FEV1).
Forced Expiratory Volume in One Second | 1 day
  a spirometer device (Minispir®, PC-based Spirometer with Oximetry option, Italy) will be used to measure the Forced Vital Capacity (FVC), Forced Expiratory Volume in One Second (FEV1).
Grip Strength | 1 day
  A handgrip dynamometer was used to measure the strength of the hand and forearm muscles (in kilograms) (Tanita Handgrip Meter, RM40, East Malaysia). The test was carried out with the elbow fully extended and the forearm in a neutral position. At 1-minute intervals, three measurements were taken on the subjects' dominant side. The participants were instructed to told the handgrip of the device tightly for 3 seconds[30]. For statistical analysis, the highest scores from three measurements were taken.
1-Repetition Maximum Strength | 1 day
  The indirect 1 repetition maximum (1RM) test is relatively simple, efficient, and safe when used and administered. The maximum repetition between 2 and 20 for any weight can be used to indirectly compute the 1RM value using the calculations. The formulas for calculating 1RM allow for weightlifting repetitions of less than 20 and a linear or curved relationship between the percentages of 1RMI. In order to determine the 1RM values of the study participants, indirect 1RM bench press, leg press, long pulley, leg extension, and overhead press were used. 1RM tests were performed using a weight machine (Technogym Selection 900).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Canli U, Aldhahi MI. The physiological and physical benefits of two types of concurrent training: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2024 Jan 2;16(1):8. doi: 10.1186/s13102-023-00798-x. PMID 38169423